CLINICAL TRIAL: NCT06846125
Title: Effect of Mindfulness Training Along With Strength Training on Psychological Rehabilitation and Knee Function Among Sprinters With Patellofemoral Pain
Brief Title: Mindfulness Training Along Strength Training Among Sprinters With Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/79018
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Patellofemoral Pain
Keywords: PFPs; Agility strength training; Strength training mindfulness training
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental)
  Interventions: Other: GROUP A: Combined Mindfulness and Strength Training
- Group B (Placebo Comparator)
  Interventions: Other: GROUP B: Strength Training Only

INTERVENTIONS:
Other: GROUP A: Combined Mindfulness and Strength Training — Week Exercises Reps x Sets 1-2 Mindfulness Training: Breathing exercises, body scans, and meditation. Strength Training: Bodyweight squats, glute bridges, calf raises. 10 x 2 3-4 Mindfulness Training: Guided visualization and mindfulness integration during exercises.
  Strength Training: Weighted squats, hamstring curls, lunges. 12 x 3 5-6 Mindfulness Training: Focus on movement awareness and posture during high-intensity drills.
  Strength Training: Single-leg squats, step-ups, resistance band lateral walks. 15 x 3 7-8 Mindfulness Training: Integration during advanced functional movements. Strength Training: Plyometric box jumps, Bulgarian split squats, deadlifts. 12 x 4
  Arms: Group A
Other: GROUP B: Strength Training Only — Week Exercises Reps x Sets 1-2 Bodyweight squats, glute bridges, calf raises. 10 x 2 3-4 Weighted squats, hamstring curls, lunges. 12 x 3 5-6 Single-leg squats, step-ups, resistance band lateral walks. 15 x 3 7-8 Plyometric box jumps, Bulgarian split squats, deadlifts. 12 x 4
  Arms: Group B

SUMMARY:
The study is to find out of the comparative Sprinting-induced patellofemoral pain syndrome (PFPS) causes physical and psychologicalal distress in athletes. While strength training has been used for physical rehabilitation, mindfulness training is a recent addition to rehabilitation science with the potential to improve both physical AND psychological protocols.

DETAILED DESCRIPTION:
Research on the effects of mindfulness and strength training on knee function in sprinters with patellofemoral pain is lacking, despite a wealth of studies on the psychological rehabilitation of athletes. The study's findings indicated that stress reduction and pain management enhance knee function. To improve the physical and psychological elements of sprinters with patellofemoral discomfort, this research assists them integrate mindfulness training with strength training. Strength training to improve knee stability and muscle balance, as well as mindfulness to lessen the psychological effects of pain and stress, can help sprinters with both the mental and physical aspects of patellofemoral pain. Research was being done on this combined approach in this specific population.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 18 to 25 years.
* Female runners.
* PFP conformation check (Single leg squat, and Eccentric step) (24)

Exclusion Criteria:

* Post-surgical condition from the past 6 months
* Chronic medical condition (cancer, COPD)
* Players addicted to any drugs or alcohol

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Baseline, Week 4, and Week 8 (Post-Intervention Assessment)
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme
Knee Range of Motion | Baseline, Week 4, and Week 8 (Post-Intervention Assessment)
  All the Ranges for Knee joint will be measured through Goniometer.
Knee Outcome Survey - Sports Activities Scale | Baseline, Week 4, and Week 8 (Post-Intervention Assessment)
  Functional Performance: Evaluated using the Knee Outcome Survey - Sports Activities Scale (SAS)

SECONDARY OUTCOMES:
Single-Leg Wall Sit Test | Baseline, Week 4, and Week 8 (Post-Intervention Assessment)
  Functional Endurance: Assessed using the Single-Leg Wall Sit Test (SLWST)
Self-Rating Anxiety Scale | Baseline, Week 4, and Week 8 (Post-Intervention Assessment)
  Psychological Well-being: Measured using the Self-Rating Anxiety Scale (SAS)

CONTACTS AND LOCATIONS:
Overall Officials: Ameena Iqbal, MS, Principal Investigator — Riphah International University
Locations (1):
- University of Lahore sports complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No